CLINICAL TRIAL: NCT03346018
Title: Observational Study: Definition of Immunologic Markers for the Differential Diagnosis Between Uveitis From Supposed Tuberculous Etiology and Sarcoidosis Uveitis
Brief Title: Immunologic Markers for the Differential Diagnosis Between Uveitis-TBC and Uveitis-SARC (TBC-SARC)
Acronym: TBC-SARC
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/0103969
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2020-07

CONDITIONS: Uveitis Tuberculous; Uveitis Sarcoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aqueous humor and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- uveitis of tuberculous etiology: Analysis of aqueous humor and plasma samples: The patients with diagnosis of uveitis of tuberculous etiology, undergone to paracentesis of anterior chamber, will can able to grant their aqueous humor and a sample of venous blood to the study of immunological markers to distinguish between uveitis of tuberculous etiology from uveitis by sarcoidosis through the analysis of the aqueous humor and the analysis of the plasma samples.
  Interventions: Diagnostic Test: Analysis of aqueous humor and plasma samples
- uveitis of suspect sarcoidosis: Analysis of aqueous humor and plasma samples:The patients with diagnosis of uveitis of suspect sarcoidosis, undergone to paracentesis of anterior chamber, will can able to grant their aqueous humor and a sample of venous blood to the study of immunological markers to distinguish between uveitis of tuberculous etiology from uveitis by sarcoidosis through the analysis of the aqueous humor and the analysis of the plasma samples.
  Interventions: Diagnostic Test: Analysis of aqueous humor and plasma samples
- uveitis of undifferentiated origin: Analysis of aqueous humor and plasma samples:The patients with diagnosis of uveitis of undifferentiated origin (tuberculosis/sarcoidosis), undergone to paracentesis of anterior chamber, will can able to grant their aqueous humor and a sample of venous blood to the study of immunological markers to distinguish between uveitis of tuberculous etiology from uveitis by sarcoidosis through the analysis of the aqueous humor and the analysis of the plasma samples.
  Interventions: Diagnostic Test: Analysis of aqueous humor and plasma samples

INTERVENTIONS:
Diagnostic Test: Analysis of aqueous humor and plasma samples — The collected samples will be analyzed as follow:
  1. Determination of the concentration of various cytokines, chemokines and groeth factors in aqueous humor and in the plasma.
  2. Analysis of the mononuclear cells ( T helper lymphocytes CD3+ and CD4+, T cytotoxic lymphocytes CD3+ CD8+, B lymphocytes CD19+, Natural killer lymphocytes CD56+ and CD3- and monocytes CD14+) present in the aqueous humor by cytofluorimetry.
  3. Evaluation of the presence of anti-human HSP70 antibodies in plasma samples by Western blot immunoprecipitation assays.
  4. Whenever possible (adequate number of cells), in vitro stimulation of mononuclear cells presence in aqueous humor with epitopes from tuberculosis mycobacterium antigens and the analysis of cytokines production in the supernatants.

SUMMARY:
Today there are no tests that allow to make a precise differential diagnosis between uveitis from presumed tuberculous origin and uveitis by sarcoidosis. Therefore, with this study, investigators aim to identify, in the aqueous humor and in the blood of participants (patients that suffering from one of these two forms of uveitis) the presence of immunologic markers that distinguish between uveitis of tuberculous etiology and uveitis by sarcoidosis.

DETAILED DESCRIPTION:
Both tuberculosis and sarcoidosis are chronic, multi-systemic and granulomatous pathologies that have very similar pulmonary and extra-pulmonary manifestations, and even in the case of ocular involvement it has been shown that many features of intraocular TB can also be found in participants with ocular sarcoidosis.

In this monocentric observational study investigators are asking to the participants with granulomatous uveitis, in which a tuberculosis or sarcoidosis origin is suspected and who will have undergo paracentesis of the anterior chamber, to grant part of the aqueous humor and a blood sample for this study.

The collected samples will be analyzed as follow:

1. Determination of the concentration of various cytokines, chemokines and growth factors in aqueous humor and in the plasma.
2. Analysis of the mononuclear cells ( T helper lymphocytes CD3+ (CD3 is the acronym of cluster of differentiation 3: a glycoprotein found on the surface of immune cells) and CD4+ ((CD4 is the acronym of cluster of differentiation 4), T cytotoxic lymphocytes CD3+ CD8+ (CD8 is the acronym of cluster of differentiation 8) , B lymphocytes CD19+ (CD19 is the acronym of cluster of differentiation 19), Natural killer lymphocytes CD56+ (CD56 is the acronym of cluster of differentiation 56) and CD3- and monocytes CD14+ (CD14 is the acronym of cluster of differentiation 14) present in the aqueous humor by cytofluorimetry.
3. Evaluation of the presence of anti-human HSP70 antibodies in plasma samples by Western blot immunoprecipitation assays.
4. Whenever possible (adequate number of cells), in vitro stimulation of mononuclear cells in aqueous humor with epitopes of tuberculosis mycobacterium antigens and the analysis of cytokines production in the supernatants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of uveitis of tuberculous etiology or patients with diagnosis of uveitis of suspect sarcoidosis or patients with diagnosis of uveitis of undifferentiated origin (tuberculosis/sarcoidosis)

Exclusion Criteria:

* Patients suffering from non-granulomatous uveitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be composed of patients who come at the Simple Dipartiental Structure of Ocular Immunology of the Reggio Emilia Hospital with diagnosis of granulomatous uveiti and to whom are diagnosed a uveitis of tuberculous etiology or uveitis of suspect sarcoidosis or uveitis of undifferentiated origin (tuberculosis/sarcoidosis).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Identify, in the aqueous humor and in the blood of patients suffering from granulomatous uveitis the presence of immunologic markers that distinguish between uveitis of tuberculous etiology and uveitis by sarcoidosis | 3 days
  The statistical analysis will based on the use of non parametric test between Group (Mann Whitney)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cimino, Principal Investigator — IRCCS/AUSL Reggio Emilia
Locations (1):
- IRCCS/AUSL Reggio Emilia Hospital, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No